CLINICAL TRIAL: NCT04758533
Title: Phase IB Clinical Trial to Assess the Safety, Tolerability, and Preliminary Efficacy of AloCELYVIR (Mesenchymal Allogenic Cells + ICOVIR-5) in Children, Adolescent and Young Adults With Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG) in Combination With Radiotherapy or Medulloblastoma in Relapse/Progression in Monotherapy
Brief Title: Clinical Trial to Assess the Safety and Efficacy of AloCELYVIR With Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG) in Combination With Radiotherapy or Medulloblastoma in Monotherapy
Acronym: AloCELYVIR
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Principal Investigator, Mrs. Laura Aranzasti, MD, Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIBHNJ-2020-01; 2020-004838-37 (EudraCT Number); 2022-502516-37-00 (EU CTIS Number)
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Medulloblastoma, Childhood, Recurrent
Keywords: Icovir-5; Mesenchymal stem cells; Medulloblastoma; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Medulloblastoma; Recurrence

STUDY DESIGN:
Intervention Model Description: Open, non-randomized, single-center Phase I clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AloCELYVIR (Experimental): Patients will received weekly infusion of AloCELYVIR during 8 weeks.
  Interventions: Biological: AloCELYVIR

INTERVENTIONS:
Biological: AloCELYVIR — Mesenchymal allogenic cells + ICOVIR-5: 500.000 cells/kg

SUMMARY:
The aim of this study is to assess the safety and efficacy of AloCELYVIR, which consist in bone marrow-derived allogenic mesenchymal stem cells infected with an oncolytic Adenovirus, ICOVIR-5. It has recently been proven that this type of cells are able of transporting oncolytic substances to tumor targets that are difficult to reach, such as medulloblastomas and gliomas, youth cancers located in the cranial cavity that have a poor prognosis and a fatal outcome. In addition, to exerting an anti-tumor action, this virus has the ability to stimulate the immune response, making the therapy even more effective. Thus, the diffuse intrinsic pontine glioma and the medulloblastoma in relapse/progression have been chosen to study the potential of this new advanced therapy through a weekly infusion for 8 weeks.

ELIGIBILITY:
INCLUSION CRITERIA COMMON TO THE TWO COHORTS

1. Patients aged 1 to 21 years.
2. Written informed consent signed by the patients legal representative and, if applicable, the minor (informed consent in patients 12 years of age or older).
3. Measurable or evaluable disease according to RANO criteria.
4. Appropriate functional status, organic function (renal, hepatic) and hematological values:

   * Lanksy and karnofsky functional status ≥50%. Patients who use a wheelchair due of tumor-associated paralysis will be considered as outpatients for functional status evaluation.
   * Haematology function:

     * Platelet count ≥75.000/µL (without support for 3 days)
     * Absolute neutrophil count (ANC) ≥500/ µL (without growth factor for 3 days)
     * Hemoglobin ≥ 8 g/dL (Transfusion allowed)
   * Liver and renal function

     * Glomerular filtration rate (GFR) (estimated by Schwartz ) >60 mL/min/1.73 m2
     * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN)
     * Transaminases (GOT and GPT) ≤3 × the upper limit of normal (ULN). ≤ 5 times ULN for patients with hepatic metastasis.
5. Patient able to comply with treatment and schedule of visits and assessments
6. Life expectancy of ≥8 weeks.
7. Appropriate contraceptive methods for sexually active males and females of childbearing age
8. Negative pregnancy test in blood or urine for females of childbearing age

INCLUSION CRITERIA COMMON TO THE COHORT A

1. Patient with new DIPG diagnosis (clinical, radiological, or histological in case a biopsy was performed before being included in the study).
2. Not having received previous treatment with radiotherapy or chemotherapy.
3. Patient able to receive radiotherapy

INCLUSION CRITERIA COMMON TO THE COHORT B

1. Patient diagnosed with relapsed and/or refractory medulloblastoma. Patients must have received at least surgery, radiation therapy and chemotherapy as part of standard treatment and have failed these treatments before they can participate in this study.
2. To be recovered to ≤ G1 from the toxic effects according to CTCAE derived from the previous treatments, excluding ototoxicity, alopecia and peripheral neurotoxicity.

EXCLUSION CRITERIA COMMON TO THE TWO COHORTS

1. Previous treatment with CELYVIR or AloCELYVIR.
2. Known active bacterial, viral, fungal or parasitic infection not controlled
3. Known active Hepatitis B or C virus or VIH infection.
4. If patients are treated with corticosteroids, they should be clinically stable and on stable or tapering doses of steroids for at least one week.
5. To be receiving another anti-cancer treatment not foreseen in this protocol or to anticipate receiving it during the patient's participation in the same concomitant with the experimental treatment.
6. Clinically significant or uncontrolled serious active and past systemic diseases that may pose an added risk to the patient

EXCLUSION CRITERIA COMMON TO THE COHORT A

1. Spontaneous massive intratumoral bleeding. Patients with postoperative bleeding (in case of biopsy or surgery) may be included in the study provided that the bleeding is controlled. The same rule applies for other postoperative complications (infection, loss of cerebrospinal fluid, absence of wound closure, subdural collection ...)
2. Patients who have previously received radiotherapy to the brain stem for another malignancy

EXCLUSION CRITERIA COMMON TO THE COHORT B

1. Washout period respect to previous treatments:

* At least two weeks since the last dose of chemotherapy. For patients receiving low-dose metronomic oral chemotherapy, this period is at least one week.
* At least four weeks since the autologous hematopoietic stem cell transplant
* At least two weeks since the last focal radiotherapy or six weeks in case of cranio-spinal radiotherapy.
* At least 2 weeks or 5 half-lifes (whichever occurs first) since the last dose of a biological or investigational treatment.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities rate (DLTs) | 1 Month
  Proportion of patients who has experienced a DLT

SECONDARY OUTCOMES:
Objective response rate | 24 Months
  Percentage of patients that achieve complete response or partial response according to RECIST 1.1 criteria
Feasibility of the combination/monotherapy | 1 Month
  Rate of patients meeting selection criteria who can receive at least one dose of AloCELYVIR
Incidence of treatment-Emergent Adverse Event | 2,5 Months
  Rate of related-AEs
Progression-free survival (PFS) | 24 Months
  Time from the date of first dose of study treatment to the date of progression or death (from ant cause).
Overall Survival (OS) | 24 Months
  Time from the date of first dose of study treatment to the date of death
Antiadenoviral humoral immune response in patients | 2,5 Months
  Anti-Adenovirus serotype 5 antibody titers
Antiadenoviral tumoral immune response in patients | 2,5 Months
  Number of CD8 antiadenovirus T-lymphocytes
Replication kinetics of Icovir-5 | 2,5 Months
  Quantification of circulating adenoviral particles

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Lassaletta Atienza, MD, Study Chair — Hospital Infantil Universitario Niño Jesús
Locations (1):
- Hospital Infantil Universitario Niño Jesús, Madrid, Spain